CLINICAL TRIAL: NCT06822465
Title: Pathobiomes in Gut of Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16494B; 5R01GM062344-23 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pseudomonas Aeruginosa
MeSH Terms: conditions — Pseudomonas Infections | interventions — In Vitro Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill Patients: All patients admitted to the burn intensive care unit (BICU), surgical intensive care unit (SICU), and the medical intensive care unit (MICU) longer than 24 hours at University of Chicago Medical Center
  Interventions: Other: P. aeruginosa using in vitro and in vivo assays

INTERVENTIONS:
Other: P. aeruginosa using in vitro and in vivo assays — This trial will entail collecting and screening stool samples obtained from critically ill patients for their virulence inducing capabilities on laboratory strains of P. aeruginosa using in vitro and in vivo assays. The investigators also plan to isolate strains of intestinal P. aeruginosa from stool samples to determine the prevalence of intestinal P. aeruginosa in a population of critically ill patients.

SUMMARY:
Despite powerful antibiotics, 50% of the intestinal tracts of critically ill surgical patients are colonized by Pseudomonas aeruginosa, whose mere presence in this site increases mortality fourfold by mechanisms that remain unknown. Many patients who survive the initial surgical trauma still succumb to multi-organ failure and septicemia secondary to an invasive nosocomial infection. The sequelae of shock, hypoxia, and parental nutrition result in injury to the intestinal mucosa, changes in gut permeability, and failure of intestinal defense mechanisms. These conditions put patients at risk for infection and multiple organ failure secondary to the translocation of enteric bacteria, initiating a systemic release of inflammatory mediators-a process that has been termed gut-derived sepsis.

Intestinal P. aeruginosa senses host factors released during stress and responds by activating its virulence gene machinery. As such, the presence of a highly activating intestinal milieu serves to induce virulence in strains of P. aeruginosa and this correlates to the severity of a patient's illness. While the host-pathogen interaction is a dynamic process, the study expects that as a patient's illness worsens or resolves over time, the "virulence-activating" properties of their intestinal milieu will change accordingly. This study will conduct a prospective observational trial in a population of critically ill patients at the Universtiy of Chicago Medical Center. This trial will entail collecting and screening stool samples obtained from critically ill patients for their virulence inducing capabilities on laboratory strains of P. aeruginosa using in vitro and in vivo assays. The study also plans to isolate strains of intestinal P. aeruginosa from stool samples to determine the prevalence of intestinal P. aeruginosa in a population of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Any ethnicity
* Age > 18 years and < 85 years

Exclusion Criteria:

* A known history of HIV/AIDS
* Active pregnancy
* Are incarcerated will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the burn intensive care unit (BICU), surgical intensive care unit (SICU), and the medical intensive care unit (MICU) longer than 24 hours at University of Chicago Medical Center and are expected to have a prolonged course of care will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
In vitro pyocyanin screening assay to determine if a stool sample has any virulence inducing ability on laboratory strains of P. aeruginosa | Through study completion, an average of 3 years
In vivo C. elegans lethality model to determine if liquid media culture "spiked" with stool sample filtrate will induce a lethal phenotype in laboratory strains of P. aeruginosa | Through study completion, an average of 3 years
PCR array analysis of known P. aeruginosa virulence genes following exposure to stool sample filtrate deemed to be highly activating by the in vitro pyocyanin assay and in vivo C. elegans lethality model. | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Alverdy, MD FACS FSIS, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Hyde Park, Illinois, United States